CLINICAL TRIAL: NCT04847440
Title: A Phase 2A Randomized, Double-blinded, Placebo-controlled, Multicenter, Dose Ranging Study of Safety and Efficacy of ATI-2173 in Combination With Tenofovir Disoproxil Fumarate in Subjects With Chronic Hepatitis B Virus Infection and in Subjects With Hepatitis D Virus Coinfection
Brief Title: A Study of Safety and Efficacy of ATI-2173 in Combination With Tenofovir Disoproxil Fumarate in Subjects With Chronic Hepatitis B Virus Infection and in Subjects With Hepatitis D Virus Coinfection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by the Sponsor
Sponsor: Antios Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANTT201
Record Dates: First submitted 2021-04-06; First posted 2021-04-19 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Hepatitis B, Chronic; Hepatitis D
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis D | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ATI-2173 and Viread (Experimental): ATI-2173 + Tenofovir disoproxil fumarate (Viread)
  Interventions: Drug: ATI-2173
- Placebo and Viread (Active Comparator): ATI-2173 Placebo + Tenofovir disoproxil fumarate
  Interventions: Drug: Viread
- ATI-2173, Viread and AB-729 (Experimental): ATI-2173 + Tenofovir disoproxil fumarate (Viread) + AB-729
  Interventions: Drug: AB-729
- Placebo, Viread and AB-729 Placebo (Active Comparator): ATI-2173 Placebo + Tenofovir disoproxil fumarate (Viread) + AB-729 Placebo
  Interventions: Drug: Viread

INTERVENTIONS:
Drug: ATI-2173 — ATI-2173 is a liver-targeted phosphoramidate prodrug of clevudine designed to enhance anti-HBV activity while decreasing systemic exposure to clevudine. It will be dosed as a capsule by mouth. Viread is a nucleotide analogue reverse transcriptase inhibitor used for chronic hepatitis B virus.
  Arms: ATI-2173 and Viread
Drug: Viread — Viread is a nucleotide analogue reverse transcriptase inhibitor used for chronic hepatitis B virus.
  Other Names: tenofovir disoproxil fumarate
  Arms: Placebo and Viread; Placebo, Viread and AB-729 Placebo
Drug: AB-729 — AB-729 is a potent, selective, subcutaneously administered, N-acetylgalactosamine (Ga1NAc)-conjugated small interfering ribonucleic acid (siRNA) inhibitor of HBV
  Arms: ATI-2173, Viread and AB-729

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multi center, dose ranging study of safety and efficacy in both volunteers with chronic hepatitis B virus infection and in volunteers with hepatitis D virus coinfection. Volunteers will be administered multiple oral doses of ATI-2173 and assessed for safety and efficacy including blood tests to show how the body metabolizes and eliminates the investigational drug as well as how the drug effects the virus infection.

ELIGIBILITY:
Inclusion Criteria:

ALL SUBJECTS:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. If female, meets one of the following criteria:

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:

      * Abstinence from heterosexual intercourse from the first study drug administration through to at least 6 months after the last dose of the study drug or until completion of the study, whichever is longer
      * Use a systemic contraceptive or an intrauterine device (with or without hormones), from at least 28 days prior to the first study drug administration through to at least 6 months after the last dose of the study drug or until completion of the study, whichever is longer, with a male condom or a diaphragm/cervical cap plus spermicide from the first study drug administration through to at least 30 days after the last dose of the study drug or until completion of the study, whichever is longer
      * Male partner vasectomized at least 6 months prior to the first study drug administration OR
   2. Male partner has had a vasectomy less than 6 months prior to dosing, and the female subject agrees to use an additional acceptable contraceptive method from the first study drug administration through to at least 6 months after the last dose of the study drug or until completion of the study, whichever is longer Or
   3. Is of non-childbearing potential, defined as surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (ie, at least 1 year without menses without an alternative medical condition prior to the first study drug administration and follicle-stimulating hormone [FSH] levels within the normal ranges for postmenopausal state of the clinical site at screening)
4. If male, meets one of the following criteria:

   1. Is able to procreate and agrees to use one of the accepted contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the last drug administration. Only for Cohort D: male subjects able to procreate must agree to use an accepted contraceptive regimen and not to donate sperm from the first study drug administration to at least 6 months after the last drug administration. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository) Or
   2. Is unable to procreate; defined as surgically sterile (ie, has undergone a vasectomy at least 6 months prior to the first study drug administration)
5. Male or female aged at least 18 years but not older than 70 years
6. Body mass index (BMI) within 18.0 kg/m2 to 35.0 kg/m2, inclusively
7. Light-, non- or ex-smoker (A light smoker is defined as someone using 10.0 nicotine units or less per day for at least 90 days prior to the first study drug administration [refer to APPENDIX 7 for conversions of nicotine usage]. An ex-smoker is defined as someone who completely stopped using nicotine products for at least 6 months prior to the first study drug administration)
8. Serum HBsAg positive at screening and at least 6 months prior to screening
9. For Cohorts A, B and E only, serum HBeAg positive and HBV DNA ≥ 20,000 IU/mL, or serum HBeAg negative and HBV DNA ≥ 2,000 IU/mL at screening
10. ALT and AST < 5 times the upper limit of normal (ULN) at screening and on the day prior to the first study drug administration (Day -1)

    SUBJECTS COINFECTED WITH CHRONIC HBV AND HDV ONLY:
11. HDV RNA in serum ≥ 500 IU/mL at screening and evidence of HDV infection (HDVAb or HDV RNA) at least 6 months prior to screening

    SUBJECTS IN COHORT D ONLY:
12. Serum HBsAg levels ≥ 100 IU/mL at screening

Exclusion Criteria:

1. Female who is lactating at screening
2. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. History of significant hypersensitivity to clevudine, tenofovir disoproxil fumarate or any related products (including excipients of ATI-2173, tenofovir disoproxil fumarate, and the placebo) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
5. Presence of clinically significant muscle disorders, myopathies or other forms of liver disease
6. Presence of any clinically significant disease, as captured in the medical history or evidence of findings on the physical examination, vital sign assessment and/or ECG assessment, and that would otherwise exclude subject from eligibility in the context of all other listed inclusion and exclusion criteria, as determined by an Investigator
7. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment
8. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
9. Any history of tuberculosis
10. Active illicit drug use including, but not limited to, cocaine, heroin and methamphetamine (the use of cannabinoids is acceptable)
11. Significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
12. Use of amiodarone in the 28 days prior to the first study drug administration
13. Presence or history of clinically significant gastrointestinal or kidney disease, or surgery that may affect drug bioavailability
14. Cirrhosis of the liver as determined by one of the following:

    * A score greater than F2 (or greater than F3 for HBV/HDV coinfected subjects) for liver fibrosis by FibroScan or FibroSure test within 6 months prior to screening or at the time of screening Or
    * A score greater than F2 (or greater than F3 for HBV/HDV coinfected subjects) on liver biopsy within 12 months prior to screening or at the time of screening
15. History of or known presence of hepatocellular carcinoma
16. Acute infection or any other clinically significant illness within 14 days of Day 1 of the study
17. History of organ transplantation
18. Presence of uncontrolled hypertension
19. Positive screening results to HIV Ag/Ab combo or hepatitis C virus tests
20. Any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
21. Inclusion in another cohort for this clinical study
22. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration
23. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
24. Donation of 500 mL or more of blood in the 56 days prior to the first study drug administration
25. Previous approved or investigational treatment for HBV or HDV, including nucleoside therapy, other than treatment by tenofovir or interferon alpha. Prior treatment with tenofovir or interferon alpha must have been discontinued at least 6 months prior to Screening.

    SUBJECTS WITH CHRONIC HBV (COHORTS A, B, AND D):
26. Positive screening results to HDV tests

    SUBJECTS IN COHORT D ONLY:
27. History of significant hypersensitivity to excipients of AB-729, any siRNAs, or antisense oligonucleotides (ASOs)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who experienced at least 1 treatment-emergent adverse event (TEAE) | Through study completion, an average of 1 year
The percentage of subjects who experienced at least one treatment emergent serious AE (SAE). | Through study completion, an average of 1 year
Percentage of subjects who experienced a treatment-emergent dose limiting toxicity (DLT) | Through study completion, an average of 1 year
Percentage of subjects who experienced at least one treatment emergent Grade 1, 2, 3, 4 or 5 laboratory abnormality | Through study completion, an average of 1 year
Percentage of subjects who discontinued study drug due to a TEAE | Through study completion, an average of 1 year
Alanine aminotransferase and aspartate aminotransferase levels versus time | Through study completion, an average of 1 year
Time to HBV viral load relapse in HBV-infected subjects | Through study completion, an average of 1 year
The reduction of HDV RNA on-treatment for HBV/HDV coinfected subjects | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
TE(max, HBV) up to Day 90 and through end of study with or without AB-729 or placebo + tenofovir | Through study completion, an average of 1 year
AUEC(HBV) up to Day 90 and through end of study with or without AB-729 of placebo + tenofovir | Through study completion, an average of 1 year
TE(max, HDV) up to Day 90 and through end of study | Through study completion, an average of 1 year
AUEC(HDV) up to Day 90 and through end of study | Through study completion, an average of 1 year
Baseline-adjusted maximal reduction in HBV DNA viral load (Emax,HBV) through 6 months after end of treatment following ATI-2173 + tenofovir (with or without AB-729) or placebo + tenofovir for 90 days in HBV-infected and HBV/HDV coinfected subjects | Through study completion at 6 months follow up
Baseline-adjusted maximal reduction in HDV RNA viral load (Emax,HDV) through 6 months after end of treatment following ATI-2173 + tenofovir or placebo + tenofovir for 90 days in HBV/HDV coinfected subjects | Through study completion at 6 months follow up
Cmax of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
Tmax of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
Ctrough of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
Ctau of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
AUC0-24 of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
T1/2 of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
RAC(Cmax) of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
RAC(AUC) of ATI-2173, clevudine, tenofovir and M1 in plasma | Through Day 120
Correlation between individual Day 90 clevudine and tenofovir Cmin and Emax,HBV or Emax, HDV of viral load | Through Day 90
Proportion of subjects with HBV SVR6 by treatment arm | Through study completion, an average of 1 year
Proportion of subjects with HDV SVR6 by treatment arm (HBV/HDV coinfected subjects only) | Through study completion, an average of 1 year
Proportion of subjects by treatment arm with HBV SVR12, SVR18, and SVR24 | Through study completion, an average of 1 year
Proportion of subjects by treatment arm with HDV SVR12, SVR18, and SVR24 (HBV/HDV coinfected subjects only) | Through study completion, an average of 1 year
Proportion of subjects by treatment arm with on-treatment ALT flares | Through Day 90
Proportion of subjects by treatment arm with off-treatment ALT flares, with no on-treatment ALT flares by treatment arm | From Day 90 through end of study, an average of 1 year
HBV DNA slope off-treatment | Through end of study, an average of 1 year
Effect on HBV pgRNA in subjects who reach SVR6 as measured by percentage of subjects by validated assay | Through end of study, an average of 1 year
HBV pgRNA at end of treatment by treatment arm | Through Day 90
Effect on HBsAg in subjects who reach HBV SVR6 as measured by percentage of subjects by validated assay | Through end of study, an average of 1 year
T(Emax,HBV) through 6 months after end of treatment following ATI-2173 + tenofovir for 90 days in HBV-infected subjects and in HBV/HDV coinfected subjects | Through end of study, an average of 1 year
AUEC(HBV) through 6 months after end of treatment following ATI-2173 + tenofovir for 90 days in HBV-infected subjects and in HBV/HDV coinfected subjects | Through end of study, an average of 1 year
T(Emax,HBV) through 6 months after end of treatment following ATI-2173 + tenofovir for 90 days in HBV/HDV coinfected subjects | Through end of study, an average of 1 year
AUEC(HDV) through 6 months after end of treatment following ATI-2173 + tenofovir for 90 days in HBV/HDV coinfected subjects | Through end of study, an average of 1 year
Change from baseline in HBsAg, HBV pgRNA, and HBcrAg at end of treatment and SVR6 in HBV-infected and in HBV/HDV coinfected subjects by treatment arm | Through end of study, an average of 1 year
Reduction from baseline in HBsAg, HBV pgRNA, and HBcrAg following ATI-2173 + tenofovir (with or without AB-729) or placebo + tenofovir for 90 days in HBV-infected and HBV/HDV coinfected subjects | Through end of study, an average of 1 year
Correlation between individual time to viral load relapse and Day 90 clevudine and/or tenofovir Cmin and AUC | Through Day 90
Correlation between SVR6 and Day 90 clevudine and/or tenofovir Cmin and AUC | Through Day 90

CONTACTS AND LOCATIONS:
Locations (2):
- Republican Clinical Hospital "Timofei Mosneaga" Arensia EM Unit, Chisinau, Republic of Moldova, Moldova
- Medical Center of Limited Liability Company "Harmoniya krasy", Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No